CLINICAL TRIAL: NCT04908033
Title: Ultra-high-frequency ECG for Prediction of Adverse Left Ventricular Remodeling in Permanent Right Ventricular Pacing
Brief Title: Ultra-high-frequency ECG for Prediction of Left Ventricular Remodeling
Status: Active, not recruiting | Type: Observational
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other); Regional Hospital Liberec (Other)
Responsible Party: Principal Investigator, Karol Curila, Principal investigator, Faculty Hospital Kralovske Vinohrady
Other Study IDs: EK-VP1421012
Record Dates: First submitted 2021-05-15; First posted 2021-06-01 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-03

CONDITIONS: RV Pacing; Negative Remodeling; Dyssynchrony; UHF-ECG; Physiological Pacing
Keywords: myocardial pacing; physiological pacing; negative remodeling; dyssynchrony; ultra-high-frequency ECG

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- myocardial pacing group: patients with the pacing lead placed into the right ventricle to obtain myocardial capture
  Interventions: Device: pacemaker implantation
- physiological pacing group: patients with the pacing lead placed into the His bundle or left bundle branch area
  Interventions: Device: pacemaker implantation

INTERVENTIONS:
Device: pacemaker implantation — pacemaker implantation

SUMMARY:
The main goal of the project is to prove that ultra-high-frequency ECG (UHF-ECG) can be used as a diagnostic tool that allows the prediction of patients susceptible to the negative effect of right ventricular myocardial pacing. The prediction will be based on the assessment of electrical dyssynchrony and local depolarization durations of left ventricular depolarization emerging during right ventricular pacing. If proved to be valid in left ventricular negative remodeling prediction, UHF-ECG-derived parameters of ventricular dyssynchrony could be used as markers allowing a lead placement optimization during an implant procedure. This information can help the operator to identify patients with the urgent need for physiological pacing (HB or LBBp) and patients in which a right ventricular myocardial pacing is sufficient and will not lead to the development of the negative left ventricular remodeling.

ELIGIBILITY:
Inclusion Criteria:

1. expectation of permanent right ventricular pacing with atrio-ventricular delay set to 150/180 ms (130/160 resp.) for sensed/paced atrial events during a follow-up,
2. a good quality of images during echocardiography,
3. willingness to attend clinical check-ups in the implanting center for at least two years.
4. life expectancy of at least 2 years

Exclusion Criteria:

1. planned cardiac surgery or transcatheter aortic valve implantation
2. hypertrophic cardiomyopathy
3. an indication for implantable cardioverter-defibrillator, biventricular implantable cardioverter-defibrillator, or biventricular pacemaker
4. active myocarditis
5. cardiac surgery or coronary revascularization in the last ten days
6. persistent/permanent atrial fibrillation during randomization
7. severe aortic stenosis
8. mitral valvular disease with an indication to intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 360 patients with an indication for permanent pacing due to permanent conduction disease of/below the AV node
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
negative remodeling prediction | 1 year from randomization
  * 5% drop in the left ventricular ejection fraction will be predicted by the duration of UHF-ECG electrical dyssynchrony parameter
  * 5% drop in the left ventricular ejection fraction will be predicted by the duration of UHF-ECG left ventricular lateral wall delay parameter
  * 5% drop in the left ventricular ejection fraction will be predicted by the duration of UHF-ECG V6d parameter
  * 10% drop in the left ventricular ejection fraction will be predicted by the duration of UHF-ECG left ventricular lateral wall delay parameter
  * 10% drop in the left ventricular ejection fraction will be predicted by the duration of UHF-ECG V6d parameter

SECONDARY OUTCOMES:
RV myocardial to physiological pacing comparison | 2 years from randomization
  left ventricular ejection fraction comparison between low risk right ventricular myocardial to physiological pacing group
UHF-ECG prediction of clinical outcome | 3 years from randomization
  occurence of death, myocardial infarction, worsening heart failure or upgrade to resynchronization therapy will be predicted by the duration of UHF-ECG electrical dyssynchrony, and/or left ventricular lateral wall delay and/or V6d parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Karol Curila, Prague, Czechia